CLINICAL TRIAL: NCT05915533
Title: Impact of the Implementation of Dance Therapy Workshops on the Quality of Life of Adults With Disabilities Institutionalized Within the Medico-social Establishments of the Univi Group: Longitudinal Intervention Study
Brief Title: Impact of the Implementation of Dance Therapy Workshops on the Quality of Life of Adults With Disabilities Institutionalized Within the Medico-social Establishments of the Univi Group
Acronym: danceworkshops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Médical Porte Verte (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-A01119-36
Record Dates: First submitted 2023-06-13; First posted 2023-06-23 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2023-06

CONDITIONS: Dance Therapy Workshop
MeSH Terms: interventions — Dance Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Before/after study (Other)
  Interventions: Other: Dance therapy

INTERVENTIONS:
Other: Dance therapy — Before/after study to measure the effects of the dance therapy activity on the quality of life of the disabled adults housed in the establishments of UNIVI group.

SUMMARY:
Dance is a multimodal activity involving motor, cognitive, sensory and sensory-motor skills as well as emotional and social skills. A growing body of research shows that the creative arts and physical exercise are able to alleviate disability, improve social interactions.

The Associative Group UNIVI wants to evaluate through this study the effects of the practice of dance on the quality of life of the disabled adults accomodates in social medical establishments of UNIVI group

DETAILED DESCRIPTION:
this research is an interventional study involving the human person of category 2 involving only minimal risks and constraints, it is multicentric and longitudinal prospective. This is a before/after study to measure the effects of the implementation of a dance therapy activity on the quality of life of the adults with disabilities housed in the 5 establishments of the univi group.

The dance therapy will be deployed in all the medico-social establishments participating in the study over a period of 12 weeks.

To do this, dance therapists will be recruited to provide these classes.

The dance-therapy will be carried out:

* in groups of 10 to 12 people who have given their informed consent,
* at least twice a week per group,
* over a period of 30 to 45 minutes maximum twice a week for 3 months. Several groups per establishment can be planned depending on the number of people who can and want to be included in the dance workshop.

  940 participant in the study will be inclued and followed at 1 month, 3 months and 6 months after the end of the dance therapy workshops.

ELIGIBILITY:
Inclusion Criteria:

* Adults with disabilities residing in medico-social establishments, including participant under guardianship or curatorship
* informed consent to participate in the study
* Participant with a minimum of language skills to understand instructions and simple questions

Exclusion Criteria:

* Contraindication to the practice of dance
* Adults with disabilities temporarily housed
* Severe cognitive and/or behavioral disorders that do not allow you to follow a dance workshop
* Permanent bed rest
* Non-affiliation to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-09-08 (Actual); Study Completion 2024-09-08 (Actual)

PRIMARY OUTCOMES:
WHOQOL-BREF scale | Eight months
  The WHOQOL-BREF has 26 questions and measures 4 domains: physical health, mental health, social relations and the environment.THE ANALYSIS IS DONE on the scores generated for each of the domains.the WHOQOL-BREF is generally recognized as a reliable and valid instrument for estimating quality of life

SECONDARY OUTCOMES:
Tinetti test: assessement of walking and balance | Eight months
  Tinetti test is an effective and reproductible tool for the assessement of the risk of falling, its administration time is approximately 5 to 10 minutes and evaluates static and dynamic balance
Get up and Go test | Eight months
  This test evaluates the transfers sitting, standing, walking and changes of direction
Time up and Go test | Eight months
  The time up and go test is the timed version of the get up and go test. The subject seated on a chair must get up, walk 3 meters in front of him, return to his chair and sit down. The score is given by the time in seconds.
  Interpretation: risk of falling if the score is greater than or equal to 21 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital La Porte Verte, Versailles, France

IPD SHARING:
Plan to Share IPD: No